CLINICAL TRIAL: NCT06283901
Title: Improving Diagnosis and Prediction of Outcome in Patients With Severe Disorders of Consciousness
Acronym: IMPROVE-DOC
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, prof. dr. Janneke Horn, prof. dr. J. Horn, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL82013.018.22
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury; Intracranial Hemorrhages; Subarachnoid Hemorrhage; Meningitis; Encephalitis; Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hemorrhages; Subarachnoid Hemorrhage; Meningitis; Encephalitis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with acute severe brain injury are usually admitted to the Intensive Care Unit. A substantial proportion of these patients will have disorders of consciousness (DOC) after interruption of sedation. It is difficult to reliably predict neurological outcome in these patients. Dependent on the extent of permanently damaged brain areas, DOC in patients with acute severe brain injury may improve or persist, eventually evolving into a minimal conscious state (MCS) or unresponsive wakefulness syndrome (UWS). These conditions are accompanied by long term severe disability. In current practice, the decision to withdraw life-sustaining support is made by interpreting the results of repeated bedside neurological examination and conventional CT-brain imaging. Reliable identification of patients with a possible good outcome, in whom treatment should not be withdrawn, is difficult. In this prospective observational cohort study we aim to identify patients with a good neurological outcome.

DETAILED DESCRIPTION:
In order to identify patients with a good neurological outcome a combination of diagnostic tests is used.

Clinical rating scales

* Simplified evaluation of consciousness scale (SECONDs) and the full outline of unresponsiveness (FOUR) score
* Once a week

Blood biomarkers

* Neuron specific enolase, neurofilament light, glial fibrillary acidic protein
* Sampling timepoints: 24h, 72h, 7 days and 14 days after brain injury
* Serum (STG-5) and plasma (EDTA-6) tubes, aliquoted (4 x 0.5ml) and stored at -80°C

EEG with reactivity testing

* Standard 21-electrode montage
* Stimuli protocol I: a set of 5 stimuli repeated 3 times

  1. Auditory: clapping in hands, 2. Auditory: calling patients name loudly, 3. Visual: passive eye opening, 4. Tactile: nasal tickle, 5. Noxious: sternal rub Each stimuli is applied for a duration of 5 seconds and an interval between stimuli of 30 seconds
* Stimuli protocol II: Cognitive-motor dissociation test

MRI-scan

* Sequences considered essential for patient care i.e.T1, T2, FLAIR, DWI/SWI
* Preferably, performed between 4-6 weeks after hospital admission

ELIGIBILITY:
Inclusion Criteria:

All patients that are admitted to the ICU with the following criteria will be eligible for inclusion:

1. Severe brain injury (GCS ≤ 8) as a result of:

   1. Traumatic brain injury
   2. Ischemic cerebrovascular accident
   3. Intracranial hemorrhage
   4. Meningo-encephalitis
   5. Subarachnoid hemorrhage
2. Age ≥ 18 years old
3. Written informed consent from legal representatives

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Absence of informed consent
* Moribund at ICU admission
* Progressive neurodegenerative disease
* Pre-admission life expectancy ≤ 6 months based on comorbidity
* GCS has been > 8 prior to inclusion
* Impossible to include within 24 hours after brain injury

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with acute severe brain injury admitted to the ICU of at least 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended | 6 months

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Radboud UMC, Nijmegen, Gelderland
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - Haaglanden MC, locatie Westeinde, The Hague, South Holland
  - UMC Groningen, Groningen